CLINICAL TRIAL: NCT01001052
Title: Relative Bioavailability of Colcrys™ (Colchicine, USP) 0.6 mg Tablets in Healthy Young and Elderly Volunteers Under Fasted Conditions
Brief Title: Relative Bioavailability of Colcrys™ 0.6 mg Tablets in Healthy Young and Elderly Volunteers Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Medical Director, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-09-1027
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Healthy; bioavailability
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colcrys™ - young subjects (18-30 yrs) (Experimental): One single dose of Colcrys™ 0.6mg taken by mouth on day 1
  Interventions: Drug: Colcrys™ (colchicine)
- Colcrys™ - elderly subjects (≥60 yrs) (Experimental): One single dose of Colcrys™ 0.6mg taken by mouth on day 1
  Interventions: Drug: Colcrys™ (colchicine)

INTERVENTIONS:
Drug: Colcrys™ (colchicine) — 0.6 mg taken by mouth on day 1
  Other Names: COLCRYS™

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of a single dose of Colcrys™ (colchicine) 0.6 mg when administered to a group of young , healthy subjects 18-30 years of age compared to a group of older, generally healthy subjects 60 years of age or older following an overnight fast.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of a single dose of Colcrys™ (colchicine) 0.6 mg when administered to a group of young, healthy subjects 18-30 years of age compared to a group of older, generally healthy subjects 60 years of age or older following an overnight fast. On study Day 1 following an overnight fast, twenty healthy, non-smoking, non-obese male and female subjects between the ages of 18 and 30 and twenty generally healthy, non-smoking, non-obese male and female subjects over 60 years of age will be administered one single dose of Colcrys™ (1 x 0.6 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of Colcrys. Blood sampling will continue on a non-confined basis at 36, 48, 60 and 72 hours post-dose. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vitals signs (temperature, respiratory rate, pulse rate and blood pressure) will be measured in the sitting position prior to dosing. Seated blood pressure and pulse will be measured at approximately 1, 3, 6 and 12 hours after dosing and prior to release from the facility. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-30 years of age or generally healthy adults over 60 years of age (elderly subjects with minor renal impairment may be allowed to participate at the discretion of the investigator), non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) of 18-30 kg/m2.

Exclusion Criteria:

* Recent participation (within 30 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* History of treatment for drug or alcohol addiction within the previous 12 months or excessive alcohol consumption during the past 12 months
* Significant history of chronic infectious disease, system disorders, organ dysfunction, especially cardiovascular disorders (angina, heart failure, irregular heartbeats, heart attack, hypertension, hypotension) stroke, renal or hepatic disorder, diabetes or bleeding disorders, gastrointestinal disease or psychiatric disorders.
* Presence of a medical condition requiring regular treatment with prescription drugs
* Subjects who have used any drugs or substances known to inhibit or induce drug-metabolizing enzymes within 30 days prior to the first dose and throughout the study
* Drug allergies or sensitivity to colchicine
* Positive test results for drugs of abuse at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darin B Brimhall, D.O., Principal Investigator — Novum

RESULTS

PARTICIPANT FLOW:
Groups:
- Colcrys™ (Colchicine) - Young Subjects (18-30 Years): All young subjects (18-30 years) received a single oral dose of Colcrys™ (1 x 0.6 mg) on Day 1 following an overnight fast of at least 10 hours.
- Colcrys™ (Colchicine) - Elderly Subjects (>60 Years): All elderly subjects (≥ 60 years)received a single oral dose of Colcrys™ (1 x 0.6 mg) on Day 1 following an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Colcrys™ (Colchicine) - Young Subjects (18-30 Years) | Colcrys™ (Colchicine) - Elderly Subjects (>60 Years)
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Colcrys™ - Young Subjects and Colcrys™ - Elderly Subjects: Colcrys™ (colchicine) - young subjects (18-30 years): All young subjects (18-30 years) received a single oral dose of Colcrys™ (1 x 0.6 mg) on Day 1 following an overnight fast of at least 10 hours.
  Colcrys™ (colchicine) - Elderly subjects (≥60 years): All elderly subjects (≥ 60 years)received a single oral dose of Colcrys™ (1 x 0.6 mg) on Day 1 following an overnight fast of at least 10 hours.
Arm/Group | Colcrys™ - Young Subjects and Colcrys™ - Elderly Subjects
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 42.32 (19.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 15
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that Colcrys™ (colchicine) reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 18, 24, 36, 48, 60 and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Colcrys™ (Colchicine) - Young Subjects (18-30 Years Old): All young subjects (18-30 years old) received a single oral dose of Colcrys™ (1 x 0.6 mg) on Day 1 following an overnight fast of at least 10 hours.
- Colcrys™ (Colchicine) - Elderly Subjects ≥ 60 Years): All older subjects (≥ 60 years old) received a single oral dose of Colcrys™ (1 x 0.6 mg) on Day 1 following an overnight fast of at least 10 hours.
Arm/Group | Colcrys™ (Colchicine) - Young Subjects (18-30 Years Old) | Colcrys™ (Colchicine) - Elderly Subjects ≥ 60 Years)
Number analyzed (Participants) | 20 | 18
ng/mL | 2.60 (0.71) | 2.56 (0.97)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)] for Colcrys™
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Colcrys™ (Colchicine) - Young Subjects (18-30 Years Old) | Colcrys™ (Colchicine) - Elderly Subjects ≥ 60 Years)
Number analyzed (Participants) | 20 | 18
ng*hr/mL | 22.39 (6.95) | 25.01 (6.92)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Colcrys™
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Colcrys™ (Colchicine) - Young Subjects (18-30 Years Old) | Colcrys™ (Colchicine) - Elderly Subjects ≥ 60 Years)
Number analyzed (Participants) | 20 | 18
ng*hr/mL | 20.14 (5.85) | 21.88 (6.22)

ADVERSE EVENTS:
Groups:
- Colcrys™ - Young Subjects (18-30 Years); Colcrys™ - Elderly Subjects (>60 Years Old): All subjects received a single dose of Colcrys™ (colchicine 1 x 0.6 mg) on Day 1 following an overnight fast.
Arm/Group | Colcrys™ - Young Subjects (18-30 Years) | Colcrys™ - Elderly Subjects (>60 Years Old)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 7/20 | 8/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colcrys™ - Young Subjects (18-30 Years) (N=20) | Colcrys™ - Elderly Subjects (>60 Years Old) (N=18)
somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 7 (7)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days